CLINICAL TRIAL: NCT06473376
Title: Comparison Between of Hegab Splint, Arthrocentesis, and Arthroscopy in Treatment of TMJ Closed Lock
Brief Title: Comparison Between Hegab Splint, Arthrocentesis, and Arthroscopy in Treatment of TMJ Closed Lock
Acronym: arthroscopy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Al-Azhar University (Other)
Responsible Party: Principal Investigator, Ayman Hegab, Prof. Ayman Hegab, Al-Azhar University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: AUAREC20200503-8
Record Dates: First submitted 2024-06-18; First posted 2024-06-25 (Actual); Last update posted 2024-06-25 (Actual); Status verified 2024-06

CONDITIONS: TMJ Disorder; TMJ Disc Disorder
MeSH Terms: conditions — Temporomandibular Joint Disorders | interventions — Arthrocentesis; Arthroscopy

STUDY DESIGN:
Intervention Model Description: The patients were randomly assigned to one of the following three groups: Group I (Control): patients treated by Hegab splint. Group II: patients treated by arthrocentesis with injection of HA/PRP mix plus Hegab splint. Group III: arthroscopy with injection of HA/PRP mix plus Hegab splint. The primary outcome variable was the change in pain using a visual analog scale, and improvement of maximum voluntary mouth opening. The secondary outcome variable was the change in joint sound. The third category of variables (age and sex) was evaluated in relation to the outcomes
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Group I (Control) (Other): Hegab TMJ splint
  Interventions: Procedure: arthrocentesis
- Group II (Other): arthrocentesis
  Interventions: Procedure: arthrocentesis
- GROUP III (Other): arthroscopy
  Interventions: Procedure: arthrocentesis

INTERVENTIONS:
Procedure: arthrocentesis — TMJ arthrocentesis and arthroscopy
  Other Names: arthroscopy

SUMMARY:
This prospective, randomized control study aimed to compare the Clinical Outcome of Hegab splint, Arthrocentesis, and Arthroscopy in treatment of TMJ closed lock. The study sample was derived from the population of patients who presented for evaluation and treatment of TMJ disorders.

DETAILED DESCRIPTION:
This prospective, randomized control study aimed to compare the Clinical Outcome of Hegab splint, Arthrocentesis, and Arthroscopy in treatment of TMJ closed lock. The study sample was derived from the population of patients who presented for evaluation and treatment of TMJ disorders. The patients were randomly assigned to one of the following three groups: Group I (Control): patients treated by Hegab splint. Group II: patients treated by arthrocentesis with injection of HA/PRP mix plus Hegab splint. Group III: arthroscopy with injection of HA/PRP mix plus Hegab splint. The primary outcome variable was the change in pain using a visual analog scale, and improvement of maximum voluntary mouth opening. The secondary outcome variable was the change in joint sound. The third category of variables (age and sex) was evaluated in relation to the outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Patients with TMJ closed lock confirmed

Exclusion Criteria:

* rheumatoid arthritis psoriatic arthritis juvenile arthritis those receiving anticoagulant therapy

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 45 (Actual)
Dates: Start 2020-01-14 (Actual); Primary Completion 2023-07-30 (Actual); Study Completion 2023-12-30 (Actual)

PRIMARY OUTCOMES:
change in pain using a visual analog scale, | one year
  The primary outcome variable was the change in pain using a visual analog scale (VAS), with 0 indicating the absence of pain and 10 indicating the worst pain possible
improvement of maximum voluntary mouth opening | one year
  improvement of maximum voluntary (non-assisted) mouth opening (MVMO) in millimetres.

CONTACTS AND LOCATIONS:
Locations (2):
- Egypt (2):
  - Al-Azhar UNIVERSITY, Cairo
  - Prof.Hegab, Cairo

IPD SHARING:
Plan to Share IPD: No